CLINICAL TRIAL: NCT05187923
Title: Computer Aided Tool for Diagnosis of Neck Masses in Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Yuhan Yang, Associate Professor, West China Hospital
Other Study IDs: HX-20211023
Record Dates: First submitted 2021-12-24; First posted 2022-01-12 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Neck Mass; Thyroglossal Duct Cysts; Branchial Cleft Anomalies; Dermoid and Epidermoid Cysts; Infantile Hemangiomas; Teratomas
MeSH Terms: conditions — Thyroglossal Cyst; Branchial Cleft Anomalies; Dermoid Cyst; Epidermal Cyst; Teratoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective cohort: The internal cohort was retrospectively enrolled in West China Hospital, Sichuan University from June 2010 and December 2020. It is a training and internal validation cohort.
  Interventions: Diagnostic Test: Artificial Intelligence Algorithm
- Prospective cohort: The same inclusion/exclusion criteria were applied for the same center prospectively. It is an external validation cohort.
  Interventions: Diagnostic Test: Artificial Intelligence Algorithm

INTERVENTIONS:
Diagnostic Test: Artificial Intelligence Algorithm — Different machine learning and deep learning computer aided strategies for model construction and validation.

SUMMARY:
The aim of this study was to evaluate the diagnostic efficacy of computer aided diagnostic tool for neck masses using machine learning and deep learning techniques on clinical information and radiological images in children.

DETAILED DESCRIPTION:
This study is a retrospective-prospective design by West China Hospital, Sichuan University, including clinical data and radiological images. A retrospective database was enrolled for patients with definite histological diagnosis and available radiological images from June 2010 and December 2020. The investigators have constructed deep learning and machine learning diagnostic models on this retrospective cohort and validated it internally. A prospective cohort would recruit patients found neck masses since January 2021. The proposed computer aided diagnostic models would also be validated in this prospective cohort externally. The aim of this study was to evaluate the diagnostic efficacy of computer aided diagnostic tool for neck masses using machine learning and deep learning techniques on clinical data and radiological images in children.

ELIGIBILITY:
Inclusion Criteria:

* Age up to 18 years old
* Receiving no treatment before diagnosis
* With written informed consent

Exclusion Criteria:

* Clinical data missing
* Unavailable radiological images
* Without written informed consent

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients who were found neck masses, and had completed clinical information and radiological images before operation, biopsy, neoadjuvant chemotherapy, and radiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The diagnostic accuracy of neck masses with AI-based screening tools in children | 1 month
  The diagnostic accuracy of neck masses with AI-based screening tools in children.

SECONDARY OUTCOMES:
The diagnostic sensitivity of neck masses with AI-based screening tools in children | 1 month
  The diagnostic sensitivity of neck masses with AI-based screening tools in children.
The diagnostic specificity of neck masses with AI-based screening tools in children | 1 month
  The diagnostic specificity of neck masses with AI-based screening tools in children.
The diagnostic positive predictive value of neck masses with AI-based screening tools in children | 1 month
  The diagnostic positive predictive value of neck masses with AI-based screening tools in children.
The diagnostic negative predictive value of neck masses with AI-based screening tools in children | 1 month
  The diagnostic negative predictive value of neck masses with AI-based screening tools in children

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No